CLINICAL TRIAL: NCT04203394
Title: Comparison of the Effects of Controlled Schroth Exercise and Home Programs on Body Symmetry, Deformity Perception and Quality of Life in Adolescent Idiopathic Scoliosis
Brief Title: Comparison of the Effects of Controlled Schroth Exercise and Home Exercise Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02.04.2018 2018/57-06
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
Keywords: Schroth exercise, conservative treatment, scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth Exercise Group (Experimental): 12 week , Exercises 1 hour, 2 times for a week with physiotherapist 20 minutes home exercise
  Interventions: Other: Schroth Exercise Group
- Home Exercise Group (Experimental): Home exercise 20 min at home Once, one hour to determine the Schroth program + teaching home exercises 20 minutes home exercise
  Interventions: Other: Home Exercise Group

INTERVENTIONS:
Other: Schroth Exercise Group — 12 week , Exercises 1 hour, 2 times for a week with physiotherapist 20 minutes home exercise
  Arms: Schroth Exercise Group
Other: Home Exercise Group — Home exercise 20 min at home Once, one hour to determine the Schroth program + teaching home exercises 20 minutes home exercise
  Arms: Home Exercise Group

SUMMARY:
The aim of this study is to compare the effects of Schroth 3D exercise method on home symmetry, trunk topography, scapula symmetry, pelvic symmetry, health related quality of life and cosmetic deformity perception in adolescents with idiopathic scoliosis

DETAILED DESCRIPTION:
Cobb angle measurement, which is accepted as the gold standard in patients with scoliosis, is a radiological measurement. However, in continuous follow-up, the search for other methods to obtain objective data that will provide a short term evaluation on the patient in determining the efficacy of conservative treatment continues.

In our study, individuals who meet the criteria will be evaluated at the beginning and end of the study. Sociodemographic features and scoliosis characteristics (Cobb angle, degree of bone maturation according to Risser, apex, vertebra rotation angle) will be recorded. Posterior Trunk Asymmetry Index (POTSI) will be used to determine body asymmetry, and topographic measurements will be performed with Artec Eva 3D Scanner and motion analysis will be performed with Biomechanical Motion Analysis Sistem (Model is BTS Smart DX100) . Individuals will evaluate their cosmetic deformities with the Walter Reed Visual Evaluation Scale. Scoliosis Research Society-22 will be used to measure quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scoliosis diagnosed and followed up by the attending physician
* 10-16 age group,
* Patients who voluntarily agreed to participate in the study
* Living in Antalya/TURKEY

Exclusion Criteria:

* Mental retardation, congenital scoliosis or spinal deformity, spinal surgery, neuromuscular disease, rheumatologic disease, tumor, cardiovascular or pulmonary disease, vertigo attack or balance problem, neurological disease
* İndividual who does not sign the consent form

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Root Mean Square(RMS) | 12 weeks
  Body right and left asymmetry will be examined.
3D Motion analysis | 12 weeks
  3D motion analysis with 4 cameras, symmetry of certain points will be evaluated during motion.
Postural Trunk Asymmetry Index (POTSI) | 12 weeks
  It is a method that allows an individual with AIS to evaluate body shape and asymmetry.
Walter Reed Visuel Assesment Scale | 12 weeks
  Walter Reed Visuel Assesment Scale (WRVAS) each aspect is shown with five levels of increasing severity of the seven type of deformity that are scored from minimum (1) to maximum (5). How individuals perceive their own cosmetic deformities and the effectiveness of treatment in improving cosmetic deformity can be evaluated
Scoliosis Research Society-22 | 12 weeks
  Scoliosis Research Society (SRS-22) is a simple and practical questionnaire specific to individuals with scoliosis. The questionnaire included pain, self-image, function / activity, mental health and treatment satisfaction. There are 22 questionnaire questions, scoring from 1 to 5. The minimum score is the worst score (22).

CONTACTS AND LOCATIONS:
Overall Officials: KADRIYE TOMBAK, Study Director — AKDENIZ UNIVERSITY PHYSICAL THERAPY
Locations (1):
- Akdeniz University Physical Therapy and Rehabilitation, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://link.springer.com/content/pdf/10.1007/s00586-021-06769-5.pdf